CLINICAL TRIAL: NCT03486964
Title: Observational Study on the Use of Incretins in Diabetic Patients: Evaluation of Metabolic Effects and Cardiovascular Events
Brief Title: Use of Incretins in Diabetic Patients
Status: Completed | Type: Observational
Sponsor: University of Pavia (Other)
Responsible Party: Principal Investigator, Giuseppe Derosa, Principal Investigator, University of Pavia
Other Study IDs: P-20180016468
Record Dates: First submitted 2018-03-27; First posted 2018-04-03 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Dipeptidyl-Peptidase IV Inhibitors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- DPP-4 plus other therapies: Patients in therapy with DPP-4 inhibitors in addition to sulfonylureas and/or biguanides and/or thiazolidinediones and/or insulin
  Interventions: Drug: DPP-4 inhibitors
- Other therapies: Patients in therapy with other hypoglycemic classes, such as sulphonylureas and/or biguanides and/or thiazolidinediones and/or insulin.

INTERVENTIONS:
Drug: DPP-4 inhibitors — Patients will be retrospectively evaluated after the addition of a DPP-4 inhibitor to previously taken anti-diabetic therapy
  Groups: DPP-4 plus other therapies

SUMMARY:
Observational, retrospective study, conducted in diabetic patients aimed to evaluate the effects on the glyco-metabolic control and on cardiovascular events of different DPP-4 inhibitors. Patients will be stratified in patients taking different DPP-4 in addition to sulfonylureas, biguanides, thiazolidinediones, insulin, compared to those in therapy with other hypoglycemic classes, such as sulphonylureas, biguanides, thiazolidinediones, insulin, alone or in combination, in primary and secondary prevention.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetic patients
* On oral hypoglycemic agents ± basal insulin
* In primary and secondary prevention

Exclusion Criteria:

- Patients with a follow-up of less than 8 years

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients in therapy with DPP-4 inhibitors in addition to sulfonylureas and/or biguanides and/or thiazolidinediones and/or insulin
Sampling Method: Probability Sample
Enrollment: 2234 (Actual)
Dates: Start 2018-03-27 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-05-30 (Actual)

PRIMARY OUTCOMES:
Glycated hemoglobin | 8 years
  Percentage
Fasting plasma glucose | 8 years
  mg/dl
Post-prandial plasma glucose | 8 years
  mg/dl

SECONDARY OUTCOMES:
Angina pectoris | 8 years
  Percentage
Extrasystoles | 8 years
  Percentage
Atrial fibrillation | 8 years
  Percentage
Fatal myocardial infarction | 8 years
  Percentage
Non-fatal myocardial infarction | 8 years
  Percentage
Heart failure | 8 years
  Percentage
Cardiovascular death | 8 years
  Percentage

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Policlinico San Matteo Foundation, Pavia, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: No